CLINICAL TRIAL: NCT01183533
Title: Safety of Intravenous Thrombolysis for Wake-up Stroke
Acronym: Wake-Up Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Sean Savitz, MD, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-10-0195
Record Dates: First submitted 2010-08-16; First posted 2010-08-17 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Ischemic Stroke
Keywords: Wake-Up Stroke; Ischemic stroke; ischemic stroke patients who wake-up with their symptoms
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- off label rt-PA used (Experimental): off label rt-PA used on all subject enrolled within 3 hours of waking with stroke symptoms at the standard of care dose.
  Interventions: Drug: Alteplase (iv t-PA)

INTERVENTIONS:
Drug: Alteplase (iv t-PA) — 0.9 mg/kg (maximum of 90 mg) IV t-PA will be administered with 10% bolus given over 1 minute, the rest given as an infusion over the remaining hour.
  Other Names: Activase®; Alteplase; tissue plasminogen activator; t-PA

SUMMARY:
The purpose is to demonstrate the safety of intravenous tissue plasminogen activator (IV t-PA) in ischemic stroke patients who present to the emergency department (ED) after awakening with the symptoms of suspected ischemic stroke.

DETAILED DESCRIPTION:
This is an open label, multi-center, safety study of acute treatment with IV alteplase in ischemic stroke patients who wake-up with their symptoms. The primary outcome of this study is the frequency of symptomatic hemorrhagic transformation evident within 24 hours of treatment with IV t-PA. Clinical improvement defined as a decrease in the National Institutes of Health Stroke Scale (NIHSS) score at 24 hours, 3 days and 90 days and modified Rankin Scale (mRS) score at 3 and 90 days. For patients that have computed tomographic angiogram (CTA) and computed tomographic perfusion (CTP), the incidence of large vessel occlusion will be quantified.

ELIGIBILITY:
Inclusion Criteria:

* Suspected acute ischemic stroke that occurred during sleep or patients who wake up with focal neurological symptoms. This includes all patients who were last known to be neurologically normal the night before,but then found upon awakening with stroke deficits. It will be considered that the last known onset time is the time when the patient was last known to be well.
* 18 to 80 years old
* NIHSS (National Institutes of Health Stroke Scale) ≤25
* Blood Pressure ≤185 mmHg systolic & ≤110 mmHg diastolic at the time of enrollment.

Treatment of higher systolic BP is permitted, prior to enrollment

* IV t-PA must be given within 3 hours of awakening from sleep
* Female patients of child-bearing potential must have a negative pregnancy test prior to enrollment

Exclusion Criteria:

* CT Exclusion Criteria: Hypodensity >1/3 middle cerebral artery (MCA) territory on non-contrast cranial CT scan or evidence of intracranial or subarachnoid hemorrhage
* Prior ischemic stroke within 3 months of the presenting event
* History of intracranial hemorrhage
* Known secured or unsecured cerebral aneurysm or vascular malformation
* Inability to control systolic BP > 185 mmHg or diastolic BP > 110 mmHg with IV anti-hypertensive medications
* Known coagulopathy or evidence of active bleeding
* Surgical procedures, biopsy, subclavian venous or arterial puncture, trauma within 14 days of the event
* Gastrointestinal or genitourinary bleeding within 14 days of the event
* Treated with IV heparin within the previous 24 hours & an abnormal (partial thromboplastin time) PTT
* Oral anticoagulants & an (international normalized ratio) INR >1.7
* Platelet count <100,000
* Venous glucose either <50 or >450
* Any patient who qualifies for this protocol should not be treated with (intra-arterial therapy) IAT If the treating physician believes a patient should undergo IAT, those patients should be identified a priori and not enrolled into this protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean I Savitz, MD, Principal Investigator — UT-Houston Health Science Center; Andrew D Barreto, MD, Principal Investigator — Study Co-PI
Locations (3):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - Swedish Medical Center, Englewood, Colorado
  - UT-Houston Health Science Center, Houston, Texas

REFERENCES:
- [Derived] Barreto AD, Fanale CV, Alexandrov AV, Gaffney KC, Vahidy FS, Nguyen CB, Sarraj A, Rahbar M, Grotta JC, Savitz SI; Wake-Up Stroke Investigators. Prospective, open-label safety study of intravenous recombinant tissue plasminogen activator in wake-up stroke. Ann Neurol. 2016 Aug;80(2):211-8. doi: 10.1002/ana.24700. Epub 2016 Jul 12. PMID 27273860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open for enrollment (began recruiting and screening for eligible patients) on July 13, 2010. The date of first enrollment was October 5, 2010 and the date of last enrollment was October 5, 2013. All patients were enrolled at one of five participating centers.
Groups:
- Off Label Rt-PA: Off label rt-PA used on all subjects enrolled within 3 hours of waking with stroke symptoms at the standard of care dose.
  Alteplase (iv t-PA): 0.9 mg/kg (maximum of 90 mg) IV t-PA will be administered with 10% bolus given over 1 minute, the rest given as an infusion over the remaining hour.
Period: Overall Study
Arm/Group | Off Label Rt-PA
Started | 40 (Between Oct 2010 and Oct 2013.)
Completed | 40 (- all pre-planned 40 patients received the study medication.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Off Label Rt-PA
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian, Non-Hispanic | 17
  Caucasian, Hispanic | 6
  African American | 16
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 40
National Institutes of Health Stroke Scale score, median (range) [Median (Full Range); unit: units on a scale] — National Institutes of Health Stroke Scale (NIHSS) score is a numerical 0-42 point scale that defines the severity of stroke deficits. It is routinely used in both the clinical assessment of patients as well as a research tool. Zero indicates a normal exam with no stroke deficits; whereas 42 indicates a severely affected individual who is comatose and unable to move their extremities. Unit of measure: "units on a scale".
  units on a scale | 6.5 [2 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Symptomatic Hemorrhagic Transformation Safety of iv Rt-PA in Wake up Stroke Patients
Description: The primary outcome of this study is the frequency of symptomatic hemorrhagic transformation evident within 24 hours of treatment with IV t-PA. Symptomatic was defined as significant clinical deterioration with at least a 4 point or more increase in the NIH Stroke scale.
Time Frame: 24 hours
Measure: Number; unit: cases.
Arm/Group | Off Label Rt-PA
Number analyzed (Participants) | 40
cases. | 0

2. Secondary Outcome: 90-day Modified Rankin Scale (mRS) Score 0 or 1
Description: Number of patients with mRS of 0 or 1 at 90 days. The mRS is a clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It has a minimum of 0 and a maximum of 6. Zero represents a patient that has no disability or residual stroke symptoms. A score of 1 is defined as: no significant disability: despite symptoms, able to carry out all usual duties and activities. The maximum score, 6, indicates death. A score of 2 is defined as slight disability: unable to perform all previous activities but able to look after own affairs without assistance; a score of 3 is defined as moderate disability: requiring some help but able to walk without assistance; a score of 4 is moderately severe disability: unable to walk without assistance and unable to attend to own bodily needs without assistance; a score of 5 is severe disability: bedridden, incontinent and requiring constant nursing care and attention.
Time Frame: 90 days
Population: ^ Note: 2 patients were not available for 90-day follow-up assessments.
Measure: Number; unit: participants
Arm/Group | Off Label Rt-PA
Number analyzed (Participants) | 38
participants | 20

3. Secondary Outcome: Mortality
Time Frame: 90 days
Population: Note: although 2 patients were not available for complete day 90 assessments, family/patient communication provided necessary mortality information.
Measure: Number; unit: participants
Arm/Group | Off Label Rt-PA
Number analyzed (Participants) | 40
participants | 2

ADVERSE EVENTS:
Time Frame: 30 days from rt-PA treatment.
Arm/Group | Off Label Rt-PA
Serious Adverse Events (participants affected / at risk) | 6/40
Other Adverse Events (participants affected / at risk) | 30/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off Label Rt-PA (N=40)
New (recurrent) Ischemic Stroke (Nervous system disorders) | 2 (2) — New, interval ischemic stroke.
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory Failure leading to Death Etiology: withdrawal of support after patient suffered from pneumonia, sepsis and respiratory failure.
Abscess (Infections and infestations) | 1 (1) — Abscess at Feeding tube site, requiring surgical bedside drainage and antibiotics.
Death (General disorders) | 1 (1) — Death from sepsis and aspiration pneumonia.
Cerebral Edema, malignant (Nervous system disorders) | 1 (1) — Malignant cerebral edema requiring decompressive hemicraniectomy.
Seizures with neurological deterioration (Nervous system disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — leading to mechanical ventilation and traceostomy.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Off Label Rt-PA (N=40)
Asymptomatic Intracranial Hemorrhage (Nervous system disorders) | 6 (6)
Orolingual Angioedema (Skin and subcutaneous tissue disorders) | 2 (2)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hypocalcemia (General disorders) | 7 (7)
Vertigo with nausea (General disorders) | 1 (1)
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fever (Infections and infestations) | 3 (3)
Hemorrhage (bleeding from ear) (Blood and lymphatic system disorders) | 1 (1)
Lung infiltrates (lower lobe) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD (chronic obstructive pulmonary disease) Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neurological Worsening (Nervous system disorders) | 1 (1)
Elevated Creatinine and/or BUN (Renal and urinary disorders) | 3 (5)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Hypertension (uncontrolled) (Vascular disorders) | 1 (1)
Deep Venous Thrombosis (Vascular disorders) | 2 (2)
Limb Ischemia (Vascular disorders) | 1 (1) — left foot
Insomnia (General disorders) | 1 (1)
Increased ESR rate (erythrocyte segmentation) (General disorders) | 1 (1)
Sore Throat (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 9 (9)
Increased INR (international normalized ratio) (Blood and lymphatic system disorders) | 4 (4)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Monocytopenia (Blood and lymphatic system disorders) | 1 (1)
Monocytosis (Blood and lymphatic system disorders) | 1 (1)
Increased PTT (partial thromboplastin time) (Blood and lymphatic system disorders) | 1 (1)
Hypoglycemia (General disorders) | 1 (1)
Hyperglycemia (General disorders) | 13 (16)
Hypokalemia (General disorders) | 3 (3)
Hyperkalemia (General disorders) | 3 (3)
Hypernatremia (General disorders) | 3 (3)
Hypomagnesemia (General disorders) | 1 (1)
Hyponatremia (General disorders) | 1 (1)
Hypermagnesemia (General disorders) | 1 (1)
Hypophosphatemia (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The single-arm / open-label design suffers from limitations such as possible bias in patient selection and outcome assessment. However, adverse events were adjudicated by the DSMB. Small trial size warrants caution; further studies are necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study PI will submit the manuscript of any proposed publication to the sponsor at least 45 days before publication, and the sponsor shall have the right to review and comment upon the publication. The sponsor shall provide any comments to investigator within 30 days of receipt of the proposed publication or presentation. At the end of the 30 day period, the PI shall be free to proceed with the publication or presentation provided he or she has complied with the sponsor's feedback.